CLINICAL TRIAL: NCT01342510
Title: The Evaluation of the Combination of Magnesium and Lidocaine for the Pretreatment of Pain That is Caused by the Injection of Propofol.
Brief Title: Combination of Magnesium and Lidocaine for the Pretreatment of Pain That is Caused by the Injection of Propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2010-0139
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: General Anesthesia; Intravenous Anesthesia
Keywords: Intravenous Anesthesia; General Anesthesia
MeSH Terms: interventions — Magnesium Sulfate; Lidocaine; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lidocaine (Experimental): Lidocaine 50 mg in a 10 cc syringe
  Interventions: Drug: Magnesium Sulfate; Drug: Lidocaine
- Magnesium (Experimental): Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe
  Interventions: Drug: Magnesium Sulfate
- Lidocaine/Magnesium (Experimental): Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe
  Interventions: Drug: Magnesium Sulfate; Drug: Lidocaine/Magnesium
- Control (Placebo Comparator): 0.9% saline in a 10 cc syringe
  Interventions: Drug: Magnesium Sulfate; Drug: Control

INTERVENTIONS:
Drug: Magnesium Sulfate — We propose studying Lidocaine 50 mg in a 10 cc syringe, Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe, 0.9% saline in a 10 cc syringe, Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe for pretreatment of propofol related pain on injection.
Drug: Lidocaine — We propose studying Lidocaine 50 mg in a 10 cc syringe, Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe, 0.9% saline in a 10 cc syringe, Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe for pretreatment of propofol related pain on injection.
  Arms: Lidocaine
Drug: Control — We propose studying Lidocaine 50 mg in a 10 cc syringe, Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe, 0.9% saline in a 10 cc syringe, Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe for pretreatment of propofol related pain on injection.
  Arms: Control
Drug: Lidocaine/Magnesium — We propose studying Lidocaine 50 mg in a 10 cc syringe, Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe, 0.9% saline in a 10 cc syringe, Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe for pretreatment of propofol related pain on injection.
  Arms: Lidocaine/Magnesium

SUMMARY:
Since the introduction of propofol into routine anesthesia practice, the phenomena of pain on injection has plagued anesthesia providers. Propofol, an unstable phenol, triggers the release of bradykinin on injection. This release causes a painful burning sensation in the patient at the site of injection. Anesthesia providers have attempted a large number of remedies to prevent this pain on injection. Previously explored ideas include injecting propofol into larger veins, warming of the hand with hot packs, and intravenous pretreatment with numerous other medications. Currently, pretreatment with lidocaine is commonly administered to prevent propofol injection pain. No studies to date have looked at the combination of lidocaine and magnesium in a single syringe for the pretreatment of pain on injection caused by propofol. In addition, the administration protocols that have been studied thus far do not mirror clinical practice at the University of Wisconsin. The investigators propose studying the use of magnesium and lidocaine in a single syringe for pretreatment of propofol related pain on injection.

DETAILED DESCRIPTION:
This study will involve little if any change from the typical induction of general anesthesia. Considering that lidocaine is routinely used for the induction of anesthesia, and that some anesthesia staff also inject magnesium prior to propofol, there will be little variation in the induction of anesthesia. Patients will be randomly assigned (by microsoft excel program providing a random number 1-4) to one of four groups:

1. Lidocaine 50 mg in a 10 cc syringe
2. Magnesium sulfate 0.25 g (2 mOsmol) in a 10 cc syringe
3. 0.9% saline in a 10 cc syringe
4. Lidocaine 50 mg and 0.25 g (2 mOsmol) magnesium sulfate in a 10 cc syringe

Study drugs will be prepared in identical syringes by the Pharmaceutical Research Center (PRC). Study personnel will receive a syringe labeled with the study number as well as a data collection sheet labeled with the study number. A 20 gauge angiocatheter will be inserted into the dorsum of the hand for IV fluids and medication administration. Subjects will be given preoperative 1-2 mg intravenous midazolam for sedation when the subject is en route to the operating room as is typically done at the discretion of the anesthesia provider caring for the patient. After instituting standard monitors and providing preoxygenation, the study drug will be injected. Twenty seconds later, 50 mg of propofol will be injected. Ten seconds after infusion of propofol, the subjects will then be asked a standard question about pain on injection "Are you having pain at your IV site?". Any behavioral signs such as facial grimacing, arm withdrawal, or tears will be noted. Pain will be assessed using a four point scale: 0=no pain, 1=mild pain (pain reported only in response to questioning and without behavioral signs), 2=moderate pain (pain reported in response to questioning and accompanied by a behavioral sign, or pain reported spontaneously without questioning), 3=severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears). Study key personnel will do these pain assessments; the behavioral signs and self-reporting of pain will be recorded separate from one another. The induction of anesthesia will then by completed with the appropriate amount of propofol. Formally assessing pain following injection is not something that is standard care but all patients are currently warned prior to injection that they may experience some warmth or burning at the site of their intravenous line.

ELIGIBILITY:
Inclusion Criteria:

* All adults American Society of Anesthesiologists (ASA) physical status 1 and 2 patients selected for general anesthesia.

Exclusion Criteria:

* age < 18 years
* allergy to local anesthetics
* end stage renal disease
* pregnancy
* prisoners
* patients requiring a rapid sequence induction
* refusal to participate and patients already participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher M Schroeder, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Johnson RA, Harper NJ, Chadwick S, Vohra A. Pain on injection of propofol. Methods of alleviation. Anaesthesia. 1990 Jun;45(6):439-42. doi: 10.1111/j.1365-2044.1990.tb14328.x. PMID 2200299
- [Result] Yull DN, Barkshire KF, Dexter T. Pretreatment with ketorolac and venous occlusion to reduce pain on injection of propofol. Anaesthesia. 2000 Mar;55(3):284-7. doi: 10.1046/j.1365-2044.2000.01320.x. PMID 10671850
- [Result] Huang YW, Buerkle H, Lee TH, Lu CY, Lin CR, Lin SH, Chou AK, Muhammad R, Yang LC. Effect of pretreatment with ketorolac on propofol injection pain. Acta Anaesthesiol Scand. 2002 Sep;46(8):1021-4. doi: 10.1034/j.1399-6576.2002.460816.x. PMID 12190806
- [Result] Ambesh SP, Dubey PK, Sinha PK. Ondansetron pretreatment to alleviate pain on propofol injection: a randomized, controlled, double-blinded study. Anesth Analg. 1999 Jul;89(1):197-9. doi: 10.1097/00000539-199907000-00035. PMID 10389803
- [Result] Apiliogullari S, Keles B, Apiliogullari B, Balasar M, Yilmaz H, Duman A. Comparison of diphenhydramine and lidocaine for prevention of pain after injection of propofol: a double-blind, placebo-controlled, randomized study. Eur J Anaesthesiol. 2007 Mar;24(3):235-8. doi: 10.1017/S026502150600202X. Epub 2007 Jan 4. PMID 17202008
- [Result] Ishiyama T, Kashimoto S, Oguchi T, Furuya A, Fukushima H, Kumazawa T. Clonidine-ephedrine combination reduces pain on injection of propofol and blunts hemodynamic stress responses during the induction sequence. J Clin Anesth. 2006 May;18(3):211-5. doi: 10.1016/j.jclinane.2005.08.005. PMID 16731324
- [Result] Saadawy I, Ertok E, Boker A. Painless injection of propofol: pretreatment with ketamine vs thiopental, meperidine, and lidocaine. Middle East J Anaesthesiol. 2007 Oct;19(3):631-44. PMID 18044291
- [Result] Asik I, Yorukoglu D, Gulay I, Tulunay M. Pain on injection of propofol: comparison of metoprolol with lidocaine. Eur J Anaesthesiol. 2003 Jun;20(6):487-9. doi: 10.1017/s0265021503000784. PMID 12803269
- [Result] Ghai B, Makkar JK, Bala I, Wig J. Effect of parecoxib pretreatment and venous occlusion on propofol injection pain: a prospective, randomized, double-blinded, placebo-controlled study. J Clin Anesth. 2010 Mar;22(2):88-92. doi: 10.1016/j.jclinane.2009.03.011. PMID 20304348
- [Result] Fujii Y, Itakura M. Comparison of lidocaine, metoclopramide, and flurbiprofen axetil for reducing pain on injection of propofol in Japanese adult surgical patients: a prospective, randomized, double-blind, parallel-group, placebo-controlled study. Clin Ther. 2008 Feb;30(2):280-6. doi: 10.1016/j.clinthera.2008.02.018. PMID 18343266 (Retraction: PMID 29724497 Clin Ther. 2018 Apr 30;:)
- [Result] Kwak KH, Ha J, Kim Y, Jeon Y. Efficacy of combination intravenous lidocaine and dexamethasone on propofol injection pain: a randomized, double-blind, prospective study in adult Korean surgical patients. Clin Ther. 2008 Jun;30(6):1113-9. doi: 10.1016/j.clinthera.2008.05.019. PMID 18640467
- [Result] Agarwal A, Ansari MF, Gupta D, Pandey R, Raza M, Singh PK, Shiopriye, Dhiraj S, Singh U. Pretreatment with thiopental for prevention of pain associated with propofol injection. Anesth Analg. 2004 Mar;98(3):683-6, table of contents. doi: 10.1213/01.ane.0000103266.73568.18. PMID 14980919
- [Result] Borazan H, Erdem TB, Kececioglu M, Otelcioglu S. Prevention of pain on injection of propofol: a comparison of lidocaine with different doses of paracetamol. Eur J Anaesthesiol. 2010 Mar;27(3):253-7. doi: 10.1097/EJA.0b013e328330eca2. PMID 19696679
- [Result] Kwak K, Kim J, Park S, Lim D, Kim S, Baek W, Jeon Y. Reduction of pain on injection of propofol: combination of pretreatment of remifentanil and premixture of lidocaine with propofol. Eur J Anaesthesiol. 2007 Sep;24(9):746-50. doi: 10.1017/S026502150600233X. Epub 2007 Jan 30. PMID 17261216
- [Result] Ayoglu H, Altunkaya H, Ozer Y, Yapakci O, Cukdar G, Ozkocak I. Does dexmedetomidine reduce the injection pain due to propofol and rocuronium? Eur J Anaesthesiol. 2007 Jun;24(6):541-5. doi: 10.1017/S0265021506002250. Epub 2007 Jan 23. PMID 17241503
- [Result] Memis D, Turan A, Karamanlioglu B, Sut N, Pamukcu Z. The use of magnesium sulfate to prevent pain on injection of propofol. Anesth Analg. 2002 Sep;95(3):606-8, table of contents. doi: 10.1097/00000539-200209000-00020. PMID 12198045
- [Result] Agarwal A, Dhiraj S, Raza M, Pandey R, Pandey CK, Singh PK, Singh U, Gupta D. Vein pretreatment with magnesium sulfate to prevent pain on injection of propofol is not justified. Can J Anaesth. 2004 Feb;51(2):130-3. doi: 10.1007/BF03018771. PMID 14766688
- [Result] Gajraj NM, Nathanson MH. Preventing pain during injection of propofol: the optimal dose of lidocaine. J Clin Anesth. 1996 Nov;8(7):575-7. doi: 10.1016/s0952-8180(96)00133-x. PMID 8910180
- [Result] Sasaki T, Okamura S, Kisara A, Ito M, Yogosawa K, Yagishita Y, Yogosawa T. Effect of lidocaine on pain caused by injection of propofol: comparison of three methods at two injection rates. J Anesth. 1999;13(1):14-6. doi: 10.1007/s005400050015. No abstract available. PMID 15235946
- [Result] Tramer MR, Glynn CJ. An evaluation of a single dose of magnesium to supplement analgesia after ambulatory surgery: randomized controlled trial. Anesth Analg. 2007 Jun;104(6):1374-9, table of contents. doi: 10.1213/01.ane.0000263416.14948.dc. PMID 17513629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 6/2011 and 10/2011.
Pre-assignment Details: 200 participants were consented. The participants were distributed between the groups as follows, 39 participants in the control group, 38 in the lidocaine group, 44 in the magnesium group, and 37 in the magnesium/lidocaine group. Participants did not receive study drug if ASA score or peripheral IV inserted was not a 20 gauge.
Period: Overall Study
Arm/Group | Lidocaine | Magnesium | Lidocaine/Magnesium | Control
Started | 50 | 50 | 50 | 50
Completed | 38 | 44 | 37 | 39
Not Completed | 12 | 6 | 13 | 11
Not completed — Protocol Violation | 12 | 6 | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Magnesium | Lidocaine/Magnesium | Control | Total
Number analyzed (Participants) | 38 | 44 | 37 | 39 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 41 | 33 | 31 | 140
  >=65 years | 3 | 3 | 4 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (15.3) | 44.4 (17.2) | 44.3 (16.2) | 45.3 (18.6) | 45.1 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 14 | 14 | 71
  Male | 16 | 23 | 23 | 25 | 87
Region of Enrollment [Number; unit: participants]
  United States | 38 | 44 | 37 | 39 | 158

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pain With Injection of Propofol
Description: Following injection of the study drug, 50 mg of propofol will be injected. Ten seconds after propofol, subjects will be asked a standard question about pain. Behavioral signs will be noted. Pain will be assessed using a four point scale: 0=no pain, 1=mild pain (pain reported only in response to questioning and without behavioral signs), 2=moderate pain (pain reported in response to questioning and a behavioral sign, or pain reported without questioning), 3=severe pain (strong vocal response or behavioral response).
Time Frame: Approximately 10 seconds following administration of propofol.
Measure: Number (95% Confidence Interval); unit: percentage of patients reporting pain
Arm/Group | Lidocaine | Magnesium | Lidocaine/Magnesium | Control
Number analyzed (Participants) | 38 | 44 | 37 | 39
percentage of patients reporting pain | 29 [17 to 45] | 57 [42 to 70] | 41 [26 to 56] | 46 [32 to 61]

2. Primary Outcome: Number of Patients With Pain Associated With Injection of Propofol.
Description: Ten seconds following injection of propofol, subjects were asked "Are you having pain at your IV site?" Any behavioral signs were noted. Injection pain was assessed using the following four point scale: 0 = no pain; 1 = mild pain (pain reported only in response to questioning and without behavioral signs); 2 = moderate pain (pain reported in response to questioning and accompanied by a behavioral sign, or pain reported spontaneously without questioning); and 3 = severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears).
Time Frame: < 1 minute.
Measure: Number; unit: participants reporting pain
Arm/Group | Lidocaine | Magnesium | Lidocaine/Magnesium | Control
Number analyzed (Participants) | 38 | 44 | 37 | 39
participants reporting pain | 11 | 25 | 15 | 18

ADVERSE EVENTS:
Time Frame: Less than one minute following injection in intravenous propofol.
Description: Injection pain was assessed using the following four point scale:0=no pain;1=mild(pain reported only in response to questioning);2=moderate(pain reported in response to questioning and accompanied by a behavioral sign, or pain reported spontaneously);and 3=severe(strong vocal response or response accompanied by strong behavioral sign).
Arm/Group | Lidocaine | Magnesium | Lidocaine/Magnesium | Control
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 11/50 | 25/50 | 15/50 | 18/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=50) | Magnesium (N=50) | Lidocaine/Magnesium (N=50) | Control (N=50)
Pain with injection of propofol (General disorders) | 11 (11) | 25 (25) | 15 (15) | 18 (18)

LIMITATIONS AND CAVEATS:
Problems with designation of ASA score differing from that given by anesthesiologist, insertion of a 20 gauge angiocatheter into the dorsum of the hand and anesthesia plan changing (general to monitored) prior to going to the operating room.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes